CLINICAL TRIAL: NCT00121420
Title: Phase II Trial of Motexafin Gadolinium With Whole Brain Radiation Therapy Followed by Stereotactic Radiosurgery Boost in the Treatment of Patients With Brain Metastases
Brief Title: Study of Motexafin Gadolinium With Whole Brain Radiation Therapy Followed by Stereotactic Radiosurgery Boost in the Treatment of Patients With Brain Metastases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-0224
Record Dates: First submitted 2005-07-14; First posted 2005-07-21 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Neoplasm Metastasis; Brain Neoplasms
Keywords: Brain Neoplasms/secondary; Brain neoplasms/radiotherapy; Brain metastasis; Neoplasm metastasis; Cranial irradiation; Radiosurgery; Lung Neoplasms; Breast Neoplasms; Kidney Neoplasms; Melanoma; Radiotherapy; Carcinoma, non-small cell lung
MeSH Terms: conditions — Neoplasm Metastasis; Brain Neoplasms; Lung Neoplasms; Breast Neoplasms; Kidney Neoplasms; Melanoma; Carcinoma, Non-Small-Cell Lung | interventions — motexafin gadolinium

INTERVENTIONS:
Drug: Motexafin gadolinium

SUMMARY:
The primary purpose of the study is to evaluate if motexafin gadolinium with whole brain radiation therapy followed by a stereotactic radiosurgery boost is a safe and effective treatment.

DETAILED DESCRIPTION:
Patients will receive three weeks of whole brain radiation therapy concurrent with daily motexafin gadolinium during weeks 2 and 3, followed by a stereotactic radiosurgery boost concurrent with motexafin gadolinium. Patients will be followed for radiologic response, neurologic progression, and neurocognitive progression.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Karnofsky performance status (KPS) ≥ 70
* Histologically confirmed malignancy with the presence of one to four intraparenchymal brain metastases
* Each patient must sign a study-specific Informed Consent form

Exclusion Criteria:

* Previous cranial radiation
* Complete resection of all known brain metastases
* Known leptomeningeal metastases
* Known liver metastases
* Clinical or radiologic evidence of progression (other than study lesion[s) within 1 month prior to enrollment
* Patients with metastases within 10 mm of the optic apparatus
* Patients with metastases in the brainstem, midbrain, pons, or medulla
* Planned chemotherapy during WBRT and/or SRS
* Uncontrolled hypertension
* Women who are pregnant or lactating

and Laboratory values as follows:

* LDH > 1.3 x upper limit of normal (ULN)
* ANC < 1500/mm3
* Platelets < 50,000/mm3
* Creatinine > 2.0 mg/dL
* AST or ALT > 3 x ULN
* Total bilirubin > 2 x ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45

PRIMARY OUTCOMES:
Rate of irreversible Grade 3 or any Grade 4 or 5 neurologic radiation toxicities occuring within 3 months following SRS boost

SECONDARY OUTCOMES:
Change in lesion size and number between screening MRI and SRS treatment -planning MRI
Time to neuroligic progression or death with evidence of neurologic progression
Time to neurocognitive progression

CONTACTS AND LOCATIONS:
Overall Officials: Minesh P Mehta, MD, Study Chair — University of Wisconsin, Madison
Locations (12):
- United States (9):
  - Phoenix, Arizona
  - Aurora, Colorado
  - Cleveland, Ohio
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Dallas, Texas
  - Houston, Texas
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Canada (3):
  - Montreal, Quebec
  - Québec, Quebec
  - Sherbrooke, Quebec

REFERENCES:
- [Background] Mehta MP, Rodrigus P, Terhaard CH, Rao A, Suh J, Roa W, Souhami L, Bezjak A, Leibenhaut M, Komaki R, Schultz C, Timmerman R, Curran W, Smith J, Phan SC, Miller RA, Renschler MF. Survival and neurologic outcomes in a randomized trial of motexafin gadolinium and whole-brain radiation therapy in brain metastases. J Clin Oncol. 2003 Jul 1;21(13):2529-36. doi: 10.1200/JCO.2003.12.122. PMID 12829672
- [Background] Evens AM. Motexafin gadolinium: a redox-active tumor selective agent for the treatment of cancer. Curr Opin Oncol. 2004 Nov;16(6):576-80. doi: 10.1097/01.cco.0000142073.29850.98. PMID 15627019
- [Background] Biaglow JE, Miller RA. The thioredoxin reductase/thioredoxin system: novel redox targets for cancer therapy. Cancer Biol Ther. 2005 Jan;4(1):6-13. doi: 10.4161/cbt.4.1.1434. Epub 2004 Jan 8. PMID 15684606
- [Background] Manon R, Hui S, Chinnaiyan P, Suh J, Chang E, Timmerman R, Phan S, Das R, Mehta M. The impact of mid-treatment MRI on defining boost volumes in the radiation treatment of glioblastoma multiforme. Technol Cancer Res Treat. 2004 Jun;3(3):303-7. doi: 10.1177/153303460400300308. PMID 15161323
- [Background] Meyers CA, Smith JA, Bezjak A, Mehta MP, Liebmann J, Illidge T, Kunkler I, Caudrelier JM, Eisenberg PD, Meerwaldt J, Siemers R, Carrie C, Gaspar LE, Curran W, Phan SC, Miller RA, Renschler MF. Neurocognitive function and progression in patients with brain metastases treated with whole-brain radiation and motexafin gadolinium: results of a randomized phase III trial. J Clin Oncol. 2004 Jan 1;22(1):157-65. doi: 10.1200/JCO.2004.05.128. PMID 14701778
- See also: National Brain Tumor Foundation — http://www.braintumor.org
- See also: Pharmacyclics — http://pharmacyclics.com